CLINICAL TRIAL: NCT05710939
Title: Comparison of the Effect of Scapular Stabilization Exercise Training on Posture and Pain in Fibromyalgia Patients
Brief Title: Effect of Scapular Stabilization Exercise Training on Posture and Pain in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, Director, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HakanPolat
Record Dates: First submitted 2023-01-18; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Fibromyalgia; Exercise, Compulsive; Pain; Postural; Defect
MeSH Terms: conditions — Fibromyalgia; Compulsive Exercise; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants' personal information is hidden
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scapular stabilization exercises (Active Comparator): scapular stabilization exercises applied to 1st group for 5 days/week for 6 weeks
  Interventions: Other: exercises
- classic shoulder exercises (Active Comparator): classic shoulder exercises applied to 1st group for 5 days/week for 6 weeks
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises

SUMMARY:
Our study was conducted to investigate the effect of scapular stabilization exercise training on cervical posture and pain in fibromyalgia. 59 patients aged 18-60 years were included in the study. The patients included in the study were diagnosed with fibromyalgia from the physical therapy outpatient clinic and individuals who did not have any other disease were included. The included individuals were divided into 2 groups by randomization method. Individuals were divided into scapula exercise therapy group (n=29) and classical exercise therapy group (n=30). Hotpack, tens and ultrasound applications were applied to both groups as conventional treatment before exercise. This protocol was applied to both groups for 6 weeks, 5 days a week. Following this protocol, classical shoulder exercises were given to the classical group and stabilization exercises were given to the scapular stabilization group. While the study designer applied the treatment, another designer applied the evaluation. The patients were evaluated for pain, cervical posture, functional status, and quality of life. pain was evaluated with a visual analog scale (vas), cervical posture was evaluated by tragus-wall distance, functional status was evaluated with fibromyalgia impact questionnaire and quality of life was evaluated with nottingam quality of life questionnaire. All evaluations were performed twice before and at the end of the treatment (6 weeks).

DETAILED DESCRIPTION:
Pain is usually seen in the scapular region in patients with fibromyalgia. We decided to do this study because we thought that there was no exercise for this area before in our study and that if it was done, improvements in pain and posture could be observed. Our study was conducted to investigate the effect of scapular stabilization exercise training on cervical posture and pain in fibromyalgia. 59 patients aged 18-60 years were included in the study. The patients included in the study were diagnosed with fibromyalgia from the physical therapy outpatient clinic and individuals who did not have any other disease were included. The included individuals were divided into 2 groups by randomization method. Individuals were divided into scapula exercise therapy group (n=29) and classical exercise therapy group (n=30). Hotpack, tens and ultrasound applications were applied to both groups as conventional treatment before exercise. This protocol was applied to both groups for 6 weeks, 5 days a week. Following this protocol, classical shoulder exercises (wand exercises, codman exercises and stretching exercises) were given to the classical group, and stabilization exercises (push-up exercises on the wall, scapular adduction, scapular elevation, rowing exercises) were given to the scapular stabilization group. While the study designer applied the treatment, another designer applied the evaluation. The patients were evaluated for pain, cervical posture, functional status, and quality of life. pain was evaluated with a visual analog scale (vas), cervical posture was evaluated by tragus-wall distance, functional status was evaluated with fibromyalgia impact questionnaire and quality of life was evaluated with nottingam quality of life questionnaire. All evaluations were performed twice before and at the end of the treatment (6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-60,
* Have not received any physical therapy and exercise therapy in the last 6 months,
* No musculoskeletal problems,
* Having no barriers to exercise therapy
* individuals were included in the study.

Exclusion Criteria:

* Individuals with psychological, cardiovascular and neurological problems,
* Female individuals with pregnancy status,
* Individuals who do not want to participate in physical therapy and exercise practices excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale ( VAS) | 6 weeks
  pain, This scale evaluates pain verbally. It questions the level of pain to the patients. It is between 0 and 10 points. O No pain, 10 means severe pain.
tragus-to-wall distance | 6 weeks
  cervical posture, This scale measures the cervical posture, the distance between the wall and the tragus in cm. The results vary from person to person, and increasing distance indicates that cervical posture has a poor prognosis.
fibromyalgia impact scale | 6 weeks
  functional status, This scale evaluates functional status. verbally questioned. scale type is survey. The questions asked are asked to give points between 0 and 3. 0 points always means 1 point often, 2 points sometimes, and 3 points never. activity, doing business, and well-being. It is stated that a high score does not affect the functional state of the disease, while a low score indicates that the disease affects the functional state. The total score range is between 0 points and 80 points.
Nottingham Health Profile | 6 weeks
  life quality,This scale evaluates quality of life. questions patients' problems with pain, social isolation, emotional reaction, physical activity, energy, and sleep. scale type is survey. Patients are asked and their answers are recorded. answers are yes or no. The total score scale is in 2 parts. The 1 section score range is between 0 and 600 points, and the 2nd section is between 0 and 7 points. A high score indicates that the quality of life is badly affected, while a low score indicates that the quality of life is not affected.

CONTACTS AND LOCATIONS:
Overall Officials: hakan Polat, Study Director — Sanko University

IPD SHARING:
Plan to Share IPD: No